CLINICAL TRIAL: NCT04897724
Title: The Clinical Performance of Direct Posterior Composite Restorations in Patients With Amelogenesis Imperfecta
Brief Title: Clinical Performance of Composites in Patients With Amelogenesis Imperfecta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neslihan Tekçe (Other)
Responsible Party: Sponsor-Investigator, Neslihan Tekçe, Associate Professor, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2014/247
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Amelogenesis Imperfecta; Dental Caries; Dental Composite
MeSH Terms: conditions — Amelogenesis Imperfecta; Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients have carious lesions in one or more surface of molars and premolars (Other): patients received direct composite restorations using a nanohybrid and a nonofil composite restorations
  Interventions: Other: dental composite

INTERVENTIONS:
Other: dental composite — clinical performance of composite restorations used for posterior teeth in patients with Amelogenesis Imperfecta

SUMMARY:
In AI patients, adhesion still remains the first option in order to achieve an early, minimally invasive intervention, and the altered enamel still represents an acceptable substrate for bonding in some AI variants. Many cases have revealed that the direct composite restorations provide satisfactory esthetic and functionality in restoring AI-affected teeth. The objective of this study was to evaluate the clinical performance of composite restorations in posterior teeth in patients afflicted with Amelogenesis Imperfecta using nanohybrid and nanofill composite materials

ELIGIBILITY:
Inclusion Criteria:

* the patient had to require treatment due to carious lesions in one or more surface of molars and premolars,
* AI diagnosis had to be made, which had to be verified clinically, and also confirmed by anamnestic family history, or clinical examination concerning Witkop's classification

Exclusion Criteria:

* patients with developmental enamel defects of other origins such as fluorosis, molar incisor hypomineralization;
* AI was associated with other oral developmental or systemic disorders, and dental abnormalities such as open-bite, deep-bite, and cross-bite;
* patients who were unable to provide their informed consent.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
Number of failed restorations evaluated according to the modified USPSH criteria in patients with occlusal restorations. | an average of 1 year
  In restorations, retention rate, color match, wear or loss of anatomic form, marginal discoloration, caries, marginal adaptation, and surface texture were scored success or failure according to modified United States Public Health Service (USPHS) criteria. According to this criteria, success restorations received Alfa (A) or Bravo (B) scores. Alfa (A) represents the ideal clinical situation; Bravo (B) is the clinically acceptable. Failed restorations received Charlie (C) or Delta (D) scores. Charlie (C) is the clinically unacceptable situations where the restorations had to be replaced; Delta (D) is the situation where the restoration is fractured, mobile or missing and needed to be replaced immediately.

IPD SHARING:
Plan to Share IPD: Undecided